CLINICAL TRIAL: NCT03099993
Title: Quantified Analysis of the Movements of the Upper Limb of Children With Hemiparesis Participating in the Stress Induced Therapy Program
Brief Title: Sensitivity of an Upper Limb Motion Analysis Protocol to Changes in Kinematics and Muscle Activity After Constraint Induced Therapy in Children With Hemiplegia
Acronym: MouvsupTCIHemi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC15_0310
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Unilateral Cerebral Palsy
Keywords: Unilateral cerebral palsy; kinematics; electromyography; constraint-induced therapy; muscle activation; upper limb; child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: Healthy volunteers (Other)
  Interventions: Other: Measurement of maximal forces of elbow pronosupination and flexion-extension
- B: Patient with heamiplegia (Other)
  Interventions: Other: Measurement of maximal forces of elbow pronosupination and flexion-extension
- C: Patient with heamiplegia and constraint induced therapy (Other): arm with constraint induced therapy (done before the protocol)
  Interventions: Other: Measurement of maximal forces of elbow pronosupination and flexion-extension

INTERVENTIONS:
Other: Measurement of maximal forces of elbow pronosupination and flexion-extension — Maximal forces of elbow pronosupination and flexion-extension will be measured with a portable dynamometer.

SUMMARY:
In France, Cerebral Palsy (CP) affects 1 in 450 births. It results from lesions of the brain, before, during, or shortly after birth. These non-progressive lesions cause muscle impairments, responsible for activity limitations. These muscle impairments include muscle stiffness, and muscle weakness. Children with Unilateral CP (UCP) have these impairments on only one side of the body. To compensate for activity limitations with their impaired arm, these children over-use their non-impaired arm. The objective of constraint-induced therapy (CIT) is to minimize this asymmetry which deteriorates mobility on the impaired side, by forcing the child to only use its impaired arm several hours a day during several weeks of therapy. It is known using clinical tests that this therapy improves the overall motor function of the impaired arm. However, the underlying mechanisms are yet unknown. An understanding of these mechanisms would suggest ways to maximize the effectiveness of this therapy, which requires a significant commitment from the child and its family. The investigaors propose in this project a quantitative and objective evaluation of the effect of CIT on the movements of the impaired arm of children with UCP. The investogators focus their analysis on muscle activation, to assess which aspect of muscle impairments is modified by CIT. To this end, the investigators will use sensors identical to those already used in clinics for the Quantified Gait Analysis of children with CP, recognized since 2006 by the Haute Autorité de Santé as providing key supplementary data in the evaluation of complex gait disorders. Results from this study will provide leads to optimize CIT. Some children could for example benefit from CIT paired with treatments to reduce muscle stiffness or to strengthen muscles

DETAILED DESCRIPTION:
Quantitative and objective evaluation of upper limb movements will take place in a motion analysis laboratory and will take place as follow:

* A clinical exam of the participant will be performed by the physician to collect maximal passive joint amplitudes with a goniometer and anatomical measures (length, circumference) of the upper limb.
* The participant will be equipped with surface electromyographic electrodes to measure the activation of his superficial muscles, and with retroreflective markers placed on anatomical landmarks of his thorax, shoulder, and arm, to measure upper limb kinematics with a 3D motion capture system composed of 8 VICON cameras.
* Maximal forces of elbow pronosupination and flexion-extension will be measured with a portable dynamometer.
* The participant will be placed on a height adjustable bench, in the center of the laboratory. He will be asked to perform upper limb movements:

  * A few movements not measured, to familiarize with the equipment;
  * Recorded movements: a trial is composed of a few consecutive cycles of a movement such as elbow flexion-extension. A trial usually last about 10seconds. A few seconds-time of rest is imposed between each trial. The required movements are the following: elbow flexion-extension, elbow pronosupination, and "hand to mouth".
* Finally, the participant will be asked to lie down on an exam table and to rest relax, in order to measure the electromyographic signal of his muscles at rest.

Duration of the protocol is about 1h30, with less than 30seconds of effort, and a few minutes of performing simple upper limb movements.

ELIGIBILITY:
Inclusion Criteria:

* Participants (excluding healthy volunteers) must have hemiparesis.
* Children must be between 6 and 17 years of age. The protocol requires a minimum concentration difficult to obtain for children under 6 years.
* Participants must be enrolled in a health insurance plan.

Exclusion Criteria:

* Inability to understand or follow instructions during 1h30.
* Physical incapacity to carry out the requested movements

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Upper limb muscle activation envelopes | 5 weeks
  Muscle activation envelopes come from electromyographic signals of upper limb muscles.
kinematics during active movements | 5 weeks
  Kinematics: angles, velocities, accelerations of the thorax, shoulder, elbow and wrist in the three anatomical plans (sagittal, frontal, transverse).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France